CLINICAL TRIAL: NCT07314099
Title: Évaluation d'Impact de l'Intervention du Breizh Fabribus Pour la création ou l'Adaptation d'Aide Technique personnalisée (BFB-IMPACT)
Brief Title: Impact Evaluation of Breizh Fabribus Intervention for Personalized Assistive Technology Creation or Adaptation
Acronym: BFB-IMPACT
Status: Recruiting | Type: Observational
Sponsor: Fondation Ildys (Other)
Responsible Party: Sponsor
Other Study IDs: RI2025_004
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Amputation; Functional Limitation; Autonomy of Older People; Handicaps Physical; Autonomy
Keywords: mobile workshop; 3D printing; laser cutting; personalized devices; user satisfaction; functionnal autonomy; disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In France, more than 14 million individuals report severe functional limitations, and nearly 5 million struggle with essential daily activities. Traditional barriers to assistive technology-high costs, lengthy funding delays, lack of information, and poorly fitting off-the-shelf solutions-frequently lead to underuse, dissatisfaction, and environmental waste The BFB-IMPACT study evaluates the real-world effectiveness of Breizh Fabribus, a mobile workshop equipped with 3D printing and laser-cutting that produces and customizes assistive devices on site for people with disabilities in Finistère, France region. This retrospective, single-center investigation includes all service recipients from January 2024 to December 2025 and measures changes in users' ability to perform targeted activities at three months post-intervention. Secondary outcomes include user satisfaction and device utilization. Data collection occurs from October 2025 to May 2026, with analysis anticipated in June 2026 and results published in the second half of 2026.

DETAILED DESCRIPTION:
The BFB-IMPACT protocol is a retrospective, mixed-methods study designed to assess Breizh Fabribus's impact on daily functioning and satisfaction among people with disabilities. All individuals who received at least one assistive device from Breizh Fabribus between January 1, 2024, and December 31, 2025, are identified via routine service records. Eligible participants and their caregivers are contacted by phone or mail and provided with study information and a consent form. Upon consent, baseline data-including demographics, medical history, and the nature of the activity difficulty-are extracted from initial request forms.

At the time of device delivery, each participant completes the Client Satisfaction Questionnaire (CSQ-8) to capture immediate feedback on device fit, usability, and co-creation experience. Three months later, participants receive a standardized follow-up questionnaire addressing: frequency of device use; changes in exposure to the originally problematic activity, rated on a five-point ordinal scale; satisfaction with device performance; and open-ended comments on barriers or facilitators. Data collection is conducted via secure online surveys or postal forms, with up to two reminders for nonresponders. An optional twelve-month follow-up is offered within the scheduled data-collection window (October 2025-May 2026) to explore longer-term durability of benefits.

The primary endpoint compares baseline and three-month follow-up scores on the activity exposure scale using paired statistical tests. Secondary analyses include trends in satisfaction scores, logistic regression to identify predictors of device adoption, and inductive content analysis of open-text feedback.

Data collection concludes in May 2026. Analysis is planned for June 2026, followed by manuscript preparation and dissemination to stakeholders in the second half of 2026. Continuous monitoring by the study coordinator ensures protocol adherence, timely follow-up, and resolution of any deviations.

ELIGIBILITY:
Inclusion Criteria:

* Any person who has received assistance from BFB for the creation or adaptation of assistive technology

Exclusion Criteria:

* objection to the use of their data
* Sollicitation but no delivery of technical assistance by BFB

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants are Finistère's habitants, and have received help and creation from BFB.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in frequency of exposure to the index activity limitation at three months post-intervention | Three months following delivery of the personalized assistive device.
  Change in the frequency with which participants encounter their initial activity limitation, measured via a standardized 5-point ordinal scale at baseline and at three months post-intervention. On this scale, 1 represents "never exposed to the activity limitation" and 5 indicates "exposed every day." Lower scores correspond to less frequent difficulty, while higher scores reflect more frequent difficulty with the targeted activity. This outcome assesses the impact of the personalized assistive device provided by Breizh Fabribus.

SECONDARY OUTCOMES:
Satisfaction with the Assistive Device | At device delivery and three months post-intervention.
  Participant satisfaction measured by the Client Satisfaction Questionnaire (CSQ-8: range 8-32, higher scores indicate greater satisfaction) at delivery and by the ESAT Satisfaction Scale (range: 0-10, higher scores indicate greater satisfaction) at three months.
Frequency of Device Use | Three months post-intervention
  Self-reported frequency of use in the targeted activity, measured using a 5-point Device Use Frequency Scale (1 = never, 5 = every day; higher values indicate more frequent use).
Barriers to Device Utilization | Three months post-intervention.
  Open-ended responses analyzed for reported barriers to use. Qualitative analysis.
Influence of Sociodemographic Factors | Three months post-intervention.
  Analysis of association between demographic characteristics and outcome measures based on CSQ-8, ESAT, and Device Use Frequency Scale.
Reasons for Requesting the Assistive Device | At baseline (device request/intake).
  Qualitative coding of motivations as reported by participants at intake.

OTHER OUTCOMES:
Satisfaction with the Assistive Device (12 Months) | Twelve months post-intervention.
  Participant satisfaction assessed using the ESAT Satisfaction Scale (range: 0-10, higher scores indicate greater satisfaction) at twelve months post-intervention.
Frequency of Device Use (12 Months) | Twelve months post-intervention.
  Self-reported frequency of use in the targeted activity, measured using the 5-point Device Use Frequency Scale (1 = never, 5 = every day; higher scores indicate more frequent use) at twelve months.
Barriers to Device Utilization (12 Months) | Twelve months post-intervention.
  Open-ended responses analyzed for reported barriers to use of the assistive device, assessed at twelve months post-intervention, qualitative data only.
Change in Exposure to Activity Limitation (12 Months) | Twelve months post-intervention.
  Change in the frequency with which participants encounter the initial activity limitation, measured via a standardized 5-point ordinal scale (1 = never, 5 = every day) at baseline and twelve months post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation ILDYS, Brest, Finistère, France